CLINICAL TRIAL: NCT05831956
Title: Taipei Medical University Shuang-Ho Hospital
Brief Title: The Efficacy and Safety of Using Collagen Patch on Anastomotic Site in Colorectal Surgery
Status: Completed | Type: Observational
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Tungcheng Chang, Chief of Colorectal Surgery, Taipei Medical University Shuang Ho Hospital
Other Study IDs: N202209004
Record Dates: First submitted 2023-04-16; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Anastomosis, Functional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Collagen group /Control group: Patients who received collagen patches on the anastomotic site during colectomy were allocated to the collagen group.
  Patients without collagen patches on the anastomotic site during colectomy were allocated to the control group.
  Interventions: Procedure: Laparoscopic colectomy

INTERVENTIONS:
Procedure: Laparoscopic colectomy — Patients who under went laparoscopic colectomy

SUMMARY:
In order to investigate the effects of collagen wound dressing on colonic anastomosis during colectomy, we conducted a retrospective cohort study. The goal of study was to determine whether the use of collagen wound dressing results in improving clinical outcomes for patients undergoing laparoscopic colectomy.

DETAILED DESCRIPTION:
Wound healing occurs in four distinct phases: hemostasis, inflammation, proliferation, and tissue remodeling. Numerous factors can influence these phases, which can be classified as either local or systemic. Local factors include infection, presence of foreign bodies, inadequate oxygenation, and other issues affecting the wound itself, while systemic factors encompass a wide range of considerations such as age, gender, presence of systemic disease, ischemia, stress, medication use, obesity, cigarette and alcohol use, nutritional status, and immunocompromised conditions.

Anastomotic healing in the colon is similar to the healing process in skin while there's still some differences. While the cellular and histological processes involved in colonic healing are well known, the pathophysiological process is not fully understood and requires further studies . Unlike skin healing, the process of patients undergoing colonic resection and anastomosis healing can only be inferred by observing certain parameters, such as amount of drainage, time to first flatus and defecation and the patient's symptoms. These parameters are used to guide the patient's recovery program. Complications such as anastomotic leakage, bleeding or stricture would lead to longer hospital stay, mortality and morbidity. The most devastating one is anastomotic leakage. Although we have found some strategies to lower the rate in colorectal surgery such as colon preparation or antibiotics administration, the leakage still bothers a lot.

Besides controlling the local and systemic factors, several biomaterial products have been designed to progress the healing. Collagen plays crucial roles in all of the four healing phases. As a result, collagen wound dressing, derived from bovine, equine, avian or porcine, has been applied in different sites of wound to promote healing. Several studies have concluded that collagen wound dressing resulted in better outcomes but limited to in vitro studies or animal based research. Pantelis D. concluded that fibrin in combination with the collagen patch can improve healing in high-risk mice that underwent colonic anastomosis surgery. Pommergaard HC. also concluded that the collagen wound dressing can lower the leakage rate in mouse colon anastomosis surgery.

Another limitation is that most studies have small sample sizes and lack of long term observation. Parker et al designed a non-randomized study and concluded that collagen wound dressing is safe and easy to apply in human colorectal surgery. Marano et al compared the complication rate of two cohorts and revealed that collagen wound dressing can lower the complication rate in the patients who underwent upper gastrointestinal surgery. As of now, it is premature to conclude that collagen wound dressing is effective in human colonic anastomosis due to the lack of human studies and larger sample size. In order to investigate the effects of collagen wound dressing on colonic anastomosis during colectomy, we conducted a retrospective cohort study. Our goal was to determine whether the use of collagen wound dressing results in improving clinical outcomes for patients undergoing laparoscopic colectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent laparoscopic colectomy.

Exclusion Criteria:

* Patients who underwent open surgery, emergent surgery, or had prior chemotherapy or concurrent chemoradiotherapy were excluded from the study

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent laparoscopic colectomy.
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Bowel function recovery | 0-30 days after colectomy
  The primary outcome measurements were the number of days until first flatus and defecation after surgery, which were recorded as the number of days from surgery to the first occurrence of each event.

CONTACTS AND LOCATIONS:
Overall Officials: Tung-Cheng Chang, MD,PhD, Study Chair — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Taipei Medical University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huang PY, Tsai MC, Kiu KT, Yen MH, Chang TC. Collagen patch cover facilitates recovery of bowel function after laparoscopic colectomy. BMC Surg. 2024 Feb 20;24(1):66. doi: 10.1186/s12893-024-02339-w. PMID 38378522